CLINICAL TRIAL: NCT02274675
Title: A Pilot Study of Robot-assisted Therapy for Post-stroke Forearm and Wrist Rehabilitation Training
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universiti Teknologi Malaysia (Other)
Collaborators: National Stroke Association of Malaysia (NASAM) (Unknown); Collaborative Research in Engineering, Science and Technology Center (CREST) (Unknown); Ministry of Higher Education (Lab2Market) (Unknown)
Responsible Party: Principal Investigator, Dr.Yeong Che Fai, Dr., Universiti Teknologi Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UTM-CR2-001
Record Dates: First submitted 2014-10-21; First posted 2014-10-24 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Stroke
Keywords: Stroke; Robot-assisted therapy; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Robot group (Experimental): Receive 0.5 hour of robot-assisted therapy for wrist and forearm and 1.5 hours of daily standard rehabilitation therapy
  Interventions: Device: Robot-assisted therapy for wrist and forearm; Other: Standard rehabilitation therapy

INTERVENTIONS:
Device: Robot-assisted therapy for wrist and forearm — Robot therapy by using a single degree reconfigurable robot to train for wrist and forearm rehabilitation training.
  Other Names: CR2-Haptic Rehabilitation Robot
Other: Standard rehabilitation therapy — Standard therapy of stroke rehabilitation including speech, physical, occupational therapies and group activities

SUMMARY:
A pilot study to assess the effectiveness of CR2-Haptic and determine the feasibility of including robotic therapy into the daily rehabilitation program.

DETAILED DESCRIPTION:
The objective of this study is to clinically assess the effectiveness of CR2-Haptic and determine the feasibility of including robotic therapy into the daily rehabilitation program, and investigate the acceptance from patients and therapists. Total of 7 patients will be recruited in this study, all the patients will receive 1.5 hours of standard therapy together with 0.5 hour of robot therapy every day. The robot therapy will be a 30 mins long session for 3 to 5 days per week over a period of six weeks. The study will include forearm pronation-supination and wrist flexion-extension training.

ELIGIBILITY:
Inclusion Criteria:

* Sub-acute and chronic stroke patients
* Able to rest comfortable in training set-up
* Mini-Mental Status Examination (MMSE) Score (>21)
* Motor Assessment Scale (Balance sitting >3)
* Modified Ashworth Scale (Wrist < 2)

Exclusion Criteria:

* Contractures in affected upper extremity which inhibit movements being tested

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yeong C Fai, PhD, Principal Investigator — Universiti Teknologi Malaysia
Locations (1):
- National Stroke Association of Malaysia (NASAM), Petaling Jaya, Kuala Lumpur, Malaysia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started on 1st June 2014 for 4 months duration in a stroke rehabilitation centre.
Period: Overall Study
Arm/Group | Robot Group
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Robot Group
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Motor Impairment of Wrist and Forearm [Mean (Standard Deviation); unit: Scores] — Motor impairment of the upper limb is measured by the means of the Fugl-Meyer Assessment Scale that are related to wrist and forearm component. The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index.
  Scores | 20.29 (4.86)
Motor Function Assessment of Hand Movement [Mean (Standard Deviation); unit: Scores] — Motor function that are related to wrist and forearm are measured using the Motor Assessment Scale. The Motor Assessment Scale (MAS) is a performance-based scale that was developed as a means of assessing everyday motor function in patients with stroke. In MAS, task 1 and 3 in the hand movement sub-component assessment were accessed (MAS-Hand), as the two task is the most related component to the tested movement. The score range = 2 and the best/worst score = 2/0 scores.
  Scores | 0.29 (0.76)
Spasticity Level of Wrist [Mean (Standard Deviation); unit: Scores] — The spasticity level of wrist is measured by using Modified Ashworth Scale. It measures resistance during passive soft-tissue stretching. This measure will only measure the wrist component, as forearm component is not included in this scale. The score range = 4 and the best/worst score = 0/4 scores.
  Scores | 1 (0.82)
Forearm's Active Range of Movement [Mean (Standard Deviation); unit: Angular degree] — Forearm's active range of motion (AROM) is a measurement to identify how far the person's joints range can move in pronation-supination by moving with their own effort.
  Angular degree | 76.29 (52.37)
Forearm's Passive Range of Motion [Mean (Standard Deviation); unit: Angular degree] — Forearm's passive range of motion (PROM) is a measurement to identify how far the person's joints range can move in pronation-supination directed by a person manually.
  Angular degree | 168.57 (12.19)
Wrist's Passive Range of Motion [Mean (Standard Deviation); unit: Angular degree] — Wrist's passive range of motion (PROM) is a measurement to identify how far the person's joints range can move in flexion-extension directed by a person manually.
  Angular degree | 121.57 (14.55)
Wrist's Active Range of Motion [Mean (Standard Deviation); unit: Angular degree] — Wrist's active range of motion (AROM) is a measurement to identify how far the person's joints range can move in by moving with their own effort.
  Angular degree | 64.14 (45.86)

OUTCOME MEASURES:

1. Primary Outcome: Motor Impairment of Wrist and Forearm
Description: Introduction: Motor impairment of the upper limb is measured by the means of the Fugl-Meyer Assessment Scale that are related to wrist and forearm component. The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index.
  Scores: With the component of upper extremity (max 4 scores), wrist (max 10 scores), passive joint motion (max 8 scores) and joint pain (max 8 scores), the total or maximum scores is the sum of all the component which is 30 and the minimum is 0. The score for a normal person is 30 scores. The higher the score indicates the better the condition of the subject.
  Procedure: The procedure is done according to the standard guideline of this assessment scale.
Time Frame: Motor impairment of wrist and forearm at week 6
Population: Stroke subjects in rehabilitation centre.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Robot Group
Number analyzed (Participants) | 7
Scores | 23.57 (6.58)

2. Secondary Outcome: Motor Function Assessment of Hand Movement
Description: Introduction: Motor function that are related to wrist and forearm are measured using the Motor Assessment Scale. The Motor Assessment Scale (MAS) is a performance-based scale that was developed as a means of assessing everyday motor function in patients with stroke. In MAS, task 1 and 3 in the hand movement sub-component assessment were accessed (MAS-Hand), as the two task is the most related component to the tested movement.
  Score: The total or maximum scores is 2, and minimum scores is 0. In this scale, the higher the score indicates the better the condition of the subject. The score for a healthy person is 2.
  Procedure: The procedure is done according to the standard guideline of this assessment scale.
Time Frame: Motor function of hand function at week 6
Population: Stroke subjects in rehabilitation centre.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Robot Group
Number analyzed (Participants) | 7
Scores | 1.14 (1.07)

3. Secondary Outcome: Spasticity Level of Wrist
Description: Introduction: The spasticity level of wrist is measured by using Modified Ashworth Scale. It measures resistance during passive soft-tissue stretching. This measure will only measure the wrist component, as forearm component is not included in this scale.
  Scoring: The total or maximum scores for the subscale is 4 and the minimum is 0 score. Higher scores indicates the higher the tone, lower score indicates less tone. 0 score indicates normal tone and no increase in tone, while 4 scores indicate affected part rigid in flexion or extension. All the scores will be summed.
  Procedure: The measuring procedure starts by holding the elbow as straight as possible at forearm pronated. Then, the patient's wrist is moved from maximum possible flexion to maximum possible extension. The test is performed up tp maximum of 3 times to avoid the influence of the effect of stretch.
Time Frame: Spasticity level of wrist at week 6
Population: Stroke subjects in rehabilitation centre.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Robot Group
Number analyzed (Participants) | 7
Scores | 0.57 (0.79)

4. Secondary Outcome: Forearm's Active Range of Movement
Description: Introduction: Forearm's active range of motion (AROM) is a measurement to identify how far the person's joints range can move in pronation-supination by moving with their own effort.
  Scores: The score is measured in terms of angular degree, where the higher the degree of motion the better the person condition. The normalized AROM for normal forearm pronation-supination is about 157 angular degree, a person who is able to achieve or over this range consider normal or in good condition in this study. The minimum angular degree will be 0.
  Procedure: The forearm AROM will be measured by using the CR2-Haptic robot, where the subject will hold the handle at forearm, subject will be guided to sit upright with shoulder abducted at 30-60' and elbow flexed at 90-120' supported by an adjustable arm rest with strap and the subject will move their forearm to maximum range in both direction. The moving range will be recorded by the robot and stored as report in its software.
Time Frame: Active range of motion of forearm at week 6
Population: Stroke subjects in rehabilitation centre.
Measure: Mean (Standard Deviation); unit: Angular degree
Arm/Group | Robot Group
Number analyzed (Participants) | 7
Angular degree | 134.71 (31.34)

5. Secondary Outcome: Forearm's Passive Range of Motion
Description: Introduction: Forearm's passive range of motion (PROM) is a measurement to identify how far the person's joints range can move in pronation-supination directed by a person manually.
  Scores: The score is measured in terms of angular degree, where the higher the degree of motion the better the person condition.The normalized forearm pronation-supination is about 169 angular degree, a person who is able to achieve or over this range is considered normal or in good condition in this study. The minimum angular degree is 0.
  Procedure: The forearm PROM will be measured by using the CR2-Haptic robot, where the subject will hold the handle at forearm, subject will be guided to sit upright with shoulder abducted at 30-60' and elbow flexed at 90-120' supported by an adjustable arm rest with strap and the forearm will be moved manually by the therapist to access the passive range of motion. The moving range will be recorded by the robot and stored as report in its software.
Time Frame: Passive range of motion of forearm at week 6
Population: Stroke subjects in rehabilitation centre.
Measure: Mean (Standard Deviation); unit: Angular degree
Arm/Group | Robot Group
Number analyzed (Participants) | 7
Angular degree | 180 (0)

6. Secondary Outcome: Wrist's Passive Range of Motion
Description: Introduction: Wrist's passive range of motion (PROM) is a measurement to identify how far the person's joints range can move in flexion-extension directed by a person manually.
  Scores: The score is measured in terms of angular degree, where the higher the degree of motion the better the person condition. The total normalized PROM for normal wrist flexion-extension is about 164 angular degree, a person who is able to achieve or over this range consider normal or in good condition in this study. The minimum angular degree is 0.
  Procedure: The wrist PROM will be measured by using the CR2-Haptic robot, where the subject will hold the handle, subject will be guided to sit upright with shoulder abducted at 30-60' and elbow flexed at 90-120' supported by an adjustable arm rest with strap and the wrist will be moved manually by the therapist to access the passive range of motion. The moving range will be recorded by the robot and store as report in its software.
Time Frame: Passive range of motion of wrist at week 6
Population: Stroke subjects in rehabilitation centre.
Measure: Mean (Standard Deviation); unit: Angular degree
Arm/Group | Robot Group
Number analyzed (Participants) | 7
Angular degree | 132 (26.39)

7. Secondary Outcome: Wrist's Active Range of Motion
Description: Introduction: Wrist's active range of motion (AROM) is a measurement to identify how far the person's joints range can move in by moving with their own effort.
  Scores: The score is measured in terms of angular degree, where the higher the degree of motion the better the person condition. The total normalized AROM for normal wrist flexion-extension is about 144 angular degree, a person who is able to achieve or over this range consider normal or in good condition in this study. The minimum angular degree is 0.
  Procedure: The wrist's AROM will be measured by using the CR2-Haptic robot, where the subject will hold the handle at forearm, subject will be guided to sit upright with shoulder abducted at 30-60' and elbow flexed at 90-120' supported by an adjustable arm rest with strap and the subject will move their wrist to maximum range in both direction. The moving range will be recorded by the robot and stored as report in its software.
Time Frame: Active range of motion of wrist at week 6
Population: Stroke subjects in rehabilitation centre.
Measure: Mean (Standard Deviation); unit: Angular degree
Arm/Group | Robot Group
Number analyzed (Participants) | 7
Angular degree | 100.14 (26.23)

ADVERSE EVENTS:
Arm/Group | Robot Group
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
The limitations of this study include the relatively small number of subjects in each group, the variation in severity level across subjects and also the lack of comparison groups to differentiate the improvement benefit from robot therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No